CLINICAL TRIAL: NCT04405466
Title: A Prospective, Epidemiological, Cohort Study to Assess the Feasibility of Screening Healthy Asymptomatic Workers for the Presence of SARS-CoV-2 by Pharyngeal Swaps and Serology at Baseline, Day 21 and Day 40
Brief Title: A Study to Assess the Feasibility of Screening for SARS-CoV-2 Among Healthy Workers
Status: Completed | Type: Observational
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: M-2020-360
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, throat swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Workers working within a production area
  Interventions: Procedure: Blood sampling; Procedure: Throat swab
- Group 2: Workers working within a laboratory area
  Interventions: Procedure: Blood sampling; Procedure: Throat swab
- Group 3: Workers working within other areas
  Interventions: Procedure: Blood sampling; Procedure: Throat swab

INTERVENTIONS:
Procedure: Blood sampling — Blood samples
Procedure: Throat swab — Throat swab

SUMMARY:
This is a prospective, epidemiological, cohort study to assess the feasibility of screening healthy asymptomatic workers for the presence of severe acute respiratory syndrome SARS-CoV-2 by pharyngeal swaps and serology at baseline, day 21 and day 40.

DETAILED DESCRIPTION:
This study has been designed to assess the feasibility of screening asymptomatic workers and to investigate the extent of infection, as determined by pharyngeal swaps analysis and immune response against the virus and virus specific CD4+ and CD8+ T-cell analysis. Furthermore, the extent to which virus-specific CD4+ and CD8+ T-cells are induced is investigated as well as the persistence of virus-specific memory CD4+ and CD8+ T-cells -especially in asymptomatic infected persons.

In total, approximately up to 500 workers will be enrolled into the trial to have 450 evaluable subjects at the end of the study. There will be three individual cohorts of workers working in different departments: workers from the production area (cohort 1), workers from the laboratory area (cohort 2) and workers working in other areas (cohort 3).

The fraction of asymptomatic or subclinical infections should be determined as well as the kinetics of the immune responses. For each timepoint the difference between the cohorts is investigated. This study also aims to evaluate the impact of sanitary and preventive measures taken within the company during the pandemic situation.

Epidemiological exposure data and biological samples will be systematically collected. The present study is being conducted in line with World Health Organization recommendations to help understanding the epidemiology of SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy workers asymptomatic for SARS-CoV-2
* Ability to consent with the study and its procedures
* Age above 18 years old
* Full time employee on site at least 3 full working days a week
* Working in a shared office/lab/manufacturing environment where at least 3 employees are present and/or having frequent contact with others i.e reception area, transportation and delivery areas.

Exclusion Criteria:

Workers presenting symptoms that could be signs of a SARS-CoV-2 infection such as:

* fever ≥38°C
* chills
* fatigue
* muscle ache (myalgia)
* sore throat
* cough
* runny nose (rhinorrhea)
* shortness of breath (dyspnea)
* wheezing
* chest pain
* other respiratory Symptoms
* headache
* nausea/vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers
Sampling Method: Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Immune responses to components of SARS-Cov-2 | up to visit 3 (day 40)
  Evaluation of immune responses to components of SARS-CoV-2 as well as evaluation of Swab for the presence of SARS-CoV-2 by PCR. Determination of the difference between the study groups in anti-SARS-CoV 2 seropositivity status. Analysis of trends in CD4/CD8 concentrations over time and correlation with immunoglobulin G (IgG) Levels and new assay evaluation.
Swabs for the presence of SARSCoV-2 | up to visit 3 (day 40)
  Evaluation of Swab for the presence of SARS-CoV-2 by PCR and determination of the difference between the study groups in anti-SARS-CoV 2 seropositivity status.

SECONDARY OUTCOMES:
Difference between the study groups in anti-SARS-CoV 2 seropositivity status | up to visit 3 (day 40)
  Evaluation of immune responses to components of SARS-CoV-2 as well as evaluation of Swab for the presence of SARS-CoV-2 by PCR. Determination of the difference between the study groups in anti-SARS-CoV 2 seropositivity status and analysis of trends in CD4/CD8 concentrations over time and correlation with IgG Levels as well as new assay evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara von Ingersleben, Dr., Principal Investigator — Miltenyi Biotec B.V. & Co. KG
Locations (1):
- Miltenyi Biotec B.V. & Co. KG, Bergisch Gladbach, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No